CLINICAL TRIAL: NCT03702933
Title: The Effects of Add-On D-serine Pharmacotherapy in Chronic Treatment Resistant Schizophrenia Patients
Brief Title: D-serine in Schizophrenia
Acronym: DSRSZ
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Herzog Hospital (Other)
Responsible Party: Principal Investigator, Heresco-Levi Uriel, Professor of Psychiatry, Herzog Hospital
Other Study IDs: HerzogHospital
Record Dates: First submitted 2018-10-09; First posted 2018-10-11 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Placebo: starch
  Interventions: Dietary Supplement: D-serine
- High Dose: 3.5 g/d D-serine adjuvant treatment
  Interventions: Dietary Supplement: D-serine
- Low Dose: 2.1 g/d D-serine adjuvant treatment
  Interventions: Dietary Supplement: D-serine

INTERVENTIONS:
Dietary Supplement: D-serine — dosage
  Other Names: placebo

SUMMARY:
This study will assess the effects of D-serine adjuvant treatment to the ongoing pharmacological treatment of schizophrenia patients that are resistant to treatments.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 Schizophrenia criteria, able and willing to give informed consent, and comply to study procedure, adequate contraception, post-menopausal or abstinent, PANSS Total Score equal or greater than 70, score of 4 or greater on two psychotic items

Exclusion Criteria:

* clinically significant, uncontrollable or unstable medical condition, mental retardation or severe organic brain syndrome, significant risk of suicide or violent behavior

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: schizophrenia patients that do not respond to their treatments
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
PANSS Total Score | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Uriel Heresco-Levy, MD, Principal Investigator — Herzog Hospital
Locations (1):
- Herzog Hospital, Jerusalem, Israel